CLINICAL TRIAL: NCT04022538
Title: Evaluation of Vertical Bone Augmentation Using Anterior Maxillary Segmental Sandwich Osteotomy: Simultaneous Versus Delayed Implant Placement, A Randomized Controlled Trial
Brief Title: Evaluation of Vertical Height in Anterior Maxillary Sandwich Osteotomy: Simultaneous Versus Delayed Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Ali Abdulkhaleq Al-dubai, Master Candidate of Oral & Maxillofacial Surgery, Faculty of Oral & Dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-05-27
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Alveolar Bone Resorption
Keywords: Vertical bone augmentation; Inlay bone graft; Dental Implants; Sandwich Osteotomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sandwich osteotomy with simultaneous implant placement (Experimental): This group will undergo Sandwich osteotomy procedure and segment will be fixed using the dental implants placed simultaneously during the same surgical procedure. The remaining gap will be filled using xenograft.
  Interventions: Procedure: Anterior maxillary vertical segmental sandwich osteotomy with simultaneous implant placement
- Sandwich osteotomy using micro-plates fixation (Active Comparator): This group will undergo Sandwich osteotomy procedure and segment will be fixed using micro-plates and screws, and the gap will be filled using xenograft.
  Interventions: Procedure: Anterior maxillary vertical segmental sandwich osteotomy using micro-plates fixation

INTERVENTIONS:
Procedure: Anterior maxillary vertical segmental sandwich osteotomy with simultaneous implant placement — Following the Sandwich Osteotomy procedure described in the study description, the following steps will be done:
  * The first implant osteotomy will be prepared and placed while a chisel is placed between the down fractured segment and the basal bone, and then the second implant will be installed.
  * The gap between the transported segment and the basal bone will be filled with xenograft particulate bone substitute.
  * Finally, periosteal scoring will be done to allow tension-free interrupted closure using 3-0 vicryl suturing material.
  Other Names: Inlay alveolar bone grafting with simultaneous implant placement
  Arms: Sandwich osteotomy with simultaneous implant placement
Procedure: Anterior maxillary vertical segmental sandwich osteotomy using micro-plates fixation — Following the Sandwich Osteotomy procedure described in the study description, the following steps will be done:
  * The created gap between the transported segment and the basal bone will be filled with xenograft particulate bone substitute.
  * The mobilized segment is to be fixed to the basal bone using micro-plates and micro-screws.
  * Finally, periosteal scoring will be done to allow tension-free interrupted closure using 3-0 vicryl suturing material.
  Arms: Sandwich osteotomy using micro-plates fixation

SUMMARY:
Vertical bone height has always presented challenge for the clinicians especially in the anterior aesthetic zone. Therefore, this trial will attempt to compare whether better vertical bone height and implant placement technique can be achieved using simultaneous implant placement with the sandwich osteotomy, which is a time saving procedure performed in a single stage surgery; when compared to using fixation plates to support the segment followed by delayed implant placement.

DETAILED DESCRIPTION:
Fixation plates are usually used to support the segmentalized bone segment during vertical bone augmentation using sandwich osteotomy and inlay bone grafting; to minimize movement of the bone segment and allow for new bone formation. Therefore, the aim of this study is to evaluate vertical bone height achieved at the anterior maxilla in vertical segmental sandwich osteotomy with simultaneous implant placement versus the same technique using fixation plates.

Description of Sandwich Osteotomy procedure to be done:

* A full thickness pyramidal flap with buccal paracrestal incision and two vertical releasing incisions slightly divergent to each other will be made. Then the mucoperiosteal flap will be reflected exposing the whole buccal cortical plate without reflection of the palatal mucosa.
* The palatal mucosa will not be reflected to avoid disturbance of blood supply to the mobilized segment for proper healing.
* With a Tungsten carbide disc - 1 mm in thickness and 10 mm in diameter - the alveolar bone will be segmented using a horizontal cut 3 to 5 mm apical to the crest of the ridge, and two lateral vertically oblique cuts 1-2 mm away from adjacent teeth roots slightly converging toward the alveolar crest or almost parallel to each other; thus creating a trapezoid-shaped bone segment pedicled on the attached palatal tissues.
* The horizontal and the two vertical cuts will then be revised using a set of graduated ridge splitting (fine chisels) osteotomes of sequential width and a light weight mallet to ensure that the surgical cuts are down to spongy bone.
* The segment will then be mobilized crestally, pedicled on the non-reflected palatal tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 20-55 years. No sex predilection.
* Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
* Edentulous anterior maxilla with vertically deficient alveolar ridge that is less than 10 mm measured from the crest of the alveolar ridge to the nasal floor.
* Normal vertical dimension with increased inter-arch space.
* The minimum number of missing teeth in the anterior maxillary alveolar ridge is two adjacent anterior teeth.

Exclusion Criteria:

* • Intra-bony lesions (e.g. cysts) or infections (e.g. abscess) that may retard the osteotomy healing.
* Previous grafting procedures in the edentulous area.
* Deficient horizontal dimensions of the alveolar ridge i.e. width is less than 5 mm.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Final Vertical Alveolar ridge height | 4 months postoperatively
  Measured in millimeters from the crest of the alveolar ridge to the floor of nasal cavity using cone-beam computed tomography

SECONDARY OUTCOMES:
Patient Satisfaction: scale from 1 to 10 | 4 months postoperatively
  Measured on a scale from 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aldubai, Principal Investigator — Master's Degree Candidate at Faculty of Dentistry, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bashutski JD, Wang HL. Common implant esthetic complications. Implant Dent. 2007 Dec;16(4):340-8. doi: 10.1097/ID.0b013e318159ca05. PMID 18091161
- [Background] Carlsson GE, Bergman B, Hedegard B. Changes in contour of the maxillary alveolar process under immediate dentures. A longitudinal clinical and x-ray cephalometric study covering 5 years. Acta Odontol Scand. 1967 Jun;25(1):45-75. doi: 10.3109/00016356709072522. No abstract available. PMID 5233859
- [Background] El Hadidy MS, Mounir M, Abou-Elfetouh A, Barakat A. Assessment of vertical ridge augmentation and labial prominence using buccal versus palatal approaches for maxillary segmental sandwich osteotomy (inlay technique): A randomized clinical trial. Clin Implant Dent Relat Res. 2018 Oct;20(5):722-728. doi: 10.1111/cid.12653. Epub 2018 Jul 18. PMID 30019829
- [Background] Esposito M, Grusovin MG, Kwan S, Worthington HV, Coulthard P. Interventions for replacing missing teeth: bone augmentation techniques for dental implant treatment. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD003607. doi: 10.1002/14651858.CD003607.pub3. PMID 18646092
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Jensen OT, Kuhlke L, Bedard JF, White D. Alveolar segmental sandwich osteotomy for anterior maxillary vertical augmentation prior to implant placement. J Oral Maxillofac Surg. 2006 Feb;64(2):290-6. doi: 10.1016/j.joms.2005.10.021. PMID 16413903
- [Background] Kahnberg KE, Nystrom E, Bartholdsson L. Combined use of bone grafts and Branemark fixtures in the treatment of severely resorbed maxillae. Int J Oral Maxillofac Implants. 1989 Winter;4(4):297-304. PMID 2639859
- [Background] Keestra JA, Barry O, Jong Ld, Wahl G. Long-term effects of vertical bone augmentation: a systematic review. J Appl Oral Sci. 2016 Jan-Feb;24(1):3-17. doi: 10.1590/1678-775720150357. PMID 27008252
- [Background] Laviv A, Jensen OT, Tarazi E, Casap N. Alveolar sandwich osteotomy in resorbed alveolar ridge for dental implants: a 4-year prospective study. J Oral Maxillofac Surg. 2014 Feb;72(2):292-303. doi: 10.1016/j.joms.2013.09.036. Epub 2013 Oct 5. PMID 24321312
- [Background] Lim G, Lin GH, Monje A, Chan HL, Wang HL. Wound Healing Complications Following Guided Bone Regeneration for Ridge Augmentation: A Systematic Review and Meta-Analysis. Int J Oral Maxillofac Implants. 2018 January/February;33(1):41-50. doi: 10.11607/jomi.5581. Epub 2017 Sep 22. PMID 28938030
- [Background] Mansour HH, Badr A, Osman AH, Atef M. Anterior maxillary sandwich osteotomy technique with simultaneous implant placement: A novel approach for management of vertical deficiency. Clin Implant Dent Relat Res. 2019 Feb;21(1):160-168. doi: 10.1111/cid.12687. Epub 2018 Nov 9. PMID 30411842
- [Background] Milinkovic I, Cordaro L. Are there specific indications for the different alveolar bone augmentation procedures for implant placement? A systematic review. Int J Oral Maxillofac Surg. 2014 May;43(5):606-25. doi: 10.1016/j.ijom.2013.12.004. Epub 2014 Jan 19. PMID 24451333
- [Background] Mounir M, Mounir S, Abou-Elfetouh A, Shaker MA. Assessment of vertical ridge augmentation in anterior aesthetic zone using onlay xenografts with titanium mesh versus the inlay bone grafting technique: A randomized clinical trial. Int J Oral Maxillofac Surg. 2017 Nov;46(11):1458-1465. doi: 10.1016/j.ijom.2017.04.021. Epub 2017 May 16. PMID 28526551
- [Background] Nkenke E, Neukam FW. Autogenous bone harvesting and grafting in advanced jaw resorption: morbidity, resorption and implant survival. Eur J Oral Implantol. 2014 Summer;7 Suppl 2:S203-17. PMID 24977256
- [Background] Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent. 1967 Jan;17(1):21-7. doi: 10.1016/0022-3913(67)90046-7. No abstract available. PMID 5224784
- [Background] Politi M, Robiony M. Localized alveolar sandwich osteotomy for vertical augmentation of the anterior maxilla. J Oral Maxillofac Surg. 1999 Nov;57(11):1380-2. doi: 10.1016/s0278-2391(99)90883-2. No abstract available. PMID 10555808
- [Background] Rachmiel A, Shilo D, Aizenbud D, Emodi O. Vertical Alveolar Distraction Osteogenesis of the Atrophic Posterior Mandible Before Dental Implant Insertion. J Oral Maxillofac Surg. 2017 Jun;75(6):1164-1175. doi: 10.1016/j.joms.2017.01.013. Epub 2017 Jan 21. PMID 28208057
- [Background] Raghoebar GM, Meijndert L, Kalk WW, Vissink A. Morbidity of mandibular bone harvesting: a comparative study. Int J Oral Maxillofac Implants. 2007 May-Jun;22(3):359-65. PMID 17622001
- [Background] Sakkas A, Wilde F, Heufelder M, Winter K, Schramm A. Autogenous bone grafts in oral implantology-is it still a "gold standard"? A consecutive review of 279 patients with 456 clinical procedures. Int J Implant Dent. 2017 Dec;3(1):23. doi: 10.1186/s40729-017-0084-4. Epub 2017 Jun 1. PMID 28573552
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Tolstunov L. Classification of the alveolar ridge width: implant-driven treatment considerations for the horizontally deficient alveolar ridges. J Oral Implantol. 2014 Jul;40 Spec No:365-70. doi: 10.1563/aaid-joi-D-14-00023. Epub 2014 Feb 27. PMID 24575743
- [Background] Rutkowski JL. Vertical Alveolar Ridge Augmentation in Implant Dentistry: A Surgical Manual and Horizontal Alveolar Ridge Augmentation in Implant Dentistry: A Surgical Manual. Tolstunov L, ed. Hoboken, NJ: John Wiley & Sons, Inc. Hoboken, New Jersey. J Oral Implantol. 2016 Dec;42(6):518. doi: 10.1563/aaid-joi-D-Review.4206. No abstract available. PMID 28002717
- [Background] Tolstunov L, Hamrick JFE, Broumand V, Shilo D, Rachmiel A. Bone Augmentation Techniques for Horizontal and Vertical Alveolar Ridge Deficiency in Oral Implantology. Oral Maxillofac Surg Clin North Am. 2019 May;31(2):163-191. doi: 10.1016/j.coms.2019.01.005. PMID 30947846